CLINICAL TRIAL: NCT01880138
Title: Effect of Animated Cartoon for Prevention of Emergence Agitation in Children Aged 1.5 - 5 yr After General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 4-2013-0192
Record Dates: First submitted 2013-06-05; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Sevoflurane Anaesthesia
Keywords: Animated cartoon, Emergence agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- watching animated cartoon (Experimental)
  Interventions: Other: watching animated cartoon before general anesthesia
- not watching animated cartoon (Placebo Comparator)
  Interventions: Other: not watching animated cartoon beofre general anaesthesia

INTERVENTIONS:
Other: watching animated cartoon before general anesthesia
  Arms: watching animated cartoon
Other: not watching animated cartoon beofre general anaesthesia
  Arms: not watching animated cartoon

SUMMARY:
Emergence agitation (EA) in children early after sevoflurane anaesthesia is a common postoperative problem, with incidence ranging up to 80%. Younger patients, particularly in the age range from 1.5 to 5 yr of age, are at increased risk of EA. Preoperative anxiety, as measured by the modified Yale Preoperative Anxiety Scale, has been shown to increase the risk of EA for each increment of 10 points in the child's state anxiety score. So, Alleviates preoperative anxiety in Children maybe decrease the incidence and severity of EA. Preschool children enjoy watching animated cartoons, and they can be immersed to animated cartoon so they become oblivious of their surroundings. Therefore, viewing an animated cartoon maybe reduce preoperative anxiety in children. This study was performed to determine effect of animated cartoon for prevention of emergence agitation in children aged 1.5 - 5 yr after general anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. pediatric patient (1.5-5yrs) scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia

Exclusion Criteria:

1. Patients with an abnormal airway, reactive airway disease, gastroesophageal reflux disease, chronic respiratory disease, or a history of an upper respiratory tract infection in the preceding 6-week period

Ages: 17 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium (PAED) Scale | (PAED) Scale changes from the moment subjects open their eyes, and every 5 minute for 24hours
  Subjects' behavior was rated in the post-anesthesia care unit (PACU) from the moment subjects opened their eyes, and every 5 minutes until discharge from the PACU. The Pediatric Anesthesia Emergence Delirium (PAED) Scale (Sikich & Lerman, 2004) was used. The scale assesses 5 behaviors (making eye contact, purposefulness of actions, awareness of surroundings, restlessness, and consolability) on a 5-point scale that ranges from 'not at all' to 'extremely'.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University College of Medicine, Seoul, Seoul, South Korea